CLINICAL TRIAL: NCT01142219
Title: A Randomized, Controlled, Double-blind Clinical Trial of L-arginine as Adjuvant Therapy for Sickle Cell Disease
Brief Title: L-Arginine and Sickle Cell Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Fundo de Incentivo à Pesquisa do Hospital de Clinicas de Porto Alegre (FIPE) (Unknown); Associação de Amigos da Hematologia (HEMOAMIGOS) (Unknown); Ajinomoto Interamericana Indústria e Comércio Ltda. (donation of L-arginine) (Unknown)
Responsible Party: Christina Matzenbacher Bittar, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-487 cep@hcpa.ufrgs.br
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; L-arginine; hemolysis; nitric oxide; pulmonary arterial hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Hemolysis; Pulmonary Arterial Hypertension | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- L-arginine (Experimental): 0.1g/kg/day for 6 months
  Interventions: Drug: L-arginine; Drug: Placebo

INTERVENTIONS:
Drug: L-arginine — L-arginine was administered orally at a dose of 0.1g/kg/day during 6 months.
Drug: Placebo — Mannitol was administered orally at a dose of 01 g/kg/day for six months.

SUMMARY:
One of the main problems in sickle cell disease is the decreased bioavailability of nitric oxide and arginine. This study was designed to assess if treating sickle cell disease patients with L-arginine would improve pulmonary arterial pressure and other aspects.

DETAILED DESCRIPTION:
This is a phase III, randomized, double-blind, placebo-controlled clinical trial with sickle cell disease patients older than 1 year of age. The patients were randomly assigned to take 0.1 g/kg/day of either L-arginine or placebo orally. Adverse events were monitored by a safety committee. The variables were assessed while patients were in remission, as part of their routine care: weight, blood pressure, full blood cell count, creatinine and dosage of methemoglobin at baseline and at each follow-up visit. Peripheral oxygen saturation (SpO2), fetal hemoglobin, lactate dehydrogenase and tricuspid regurgitant jet velocity were measured through transthoracic Doppler echocardiogram before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle cell disease confirmed through hemoglobin electrophoresis
* Genotypes SS, SC and Sβ thalassemia
* Age > 1 year

Exclusion Criteria:

* Liver dysfunction (alanine aminotransferase ALT > 3 times the normal levels
* Renal dysfunction (creatinine > twice the normal levels)
* Increase in methemoglobin levels (> 5 times the normal levels)
* History of recent stroke (< 1 month) and priapism
* Pregnancy
* Allergy to L-arginine
* Use of sildenafil, calcium channel blockers, nitroglycerin or other nitrates

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Tricuspid regurgitant jet velocity >2.5 m/s | 6 months
  Tricuspid regurgitant jet velocity was used to assess pulmonary arterial hypertension before and after treatment with L-arginine.

SECONDARY OUTCOMES:
Lactate dehydrogenase levels | 6 months
  The effect of L-argigine administration on hemolysis was assessed through the variation of serum levels of lactate dehydrogenase.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil